CLINICAL TRIAL: NCT02049671
Title: Elucidation of the Effects of Growth Hormone (GH) Deficiency and GH Replacement on Clot and Platelet
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ED12/10391; 13/YH/0061 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-01-20; First posted 2014-01-30 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Hypopituitary Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Growth Hormone Therapy
  Interventions: Drug: Growth Hormone Therapy
- Control Group

INTERVENTIONS:
Drug: Growth Hormone Therapy
  Groups: Growth Hormone Therapy

SUMMARY:
Large population studies of hypopituitary adults (patients with pituitary gland failure) on conventional hormone replacement, but not growth hormone, have an approximate two fold increase in death rate (mortality). The vast majority of this excess mortality relates to vascular disease. While it is possible that overreplacement with steroids, underreplacement with thyroid hormones and sex hormone deficiency contribute, there are increasing data to support a role for GH in the cause of the excess vascular risk. Although a number of surrogates of vascular risk are described in patients with GH deficiency (GHD), how these translate mechanistically into atherothrombotic (blockage of the arteries) disease has not been fully elucidated.

This proposed study will analyse both traditional (body composition, serum lipids, handling of sugars)and more complex markers (inflammation, procoagulation, fibrinolysis) of vascular risk/disease. In addition the study will examine 24hr blood pressure, arterial wall thickness, clot structure and function, as well as platelet action. Measurements will be performed at baseline and will be reassessed after patients have been on a stable dose of GH replacement for at least three months.

The results of the study will characterise risk factors for vascular disease, and take this a step further to elucidate how these changes translate mechanistically in to vascular damage.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written consent
* Adults with confirmed GHD (Insulin stimulation test <3ug/L)
* Other hormone replacement therapy stable for at least three months

Exclusion Criteria:

* active malignancy
* an acute vascular event within three months of the study
* any therapy other than hormone replacement
* serum creatinine >120 micromol/l
* abnormal LFTs (ALT>3 fold upper limit of normal)

Ages: 16 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Hypopituitary adults
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-06-01 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Turbidity analysis. | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom